CLINICAL TRIAL: NCT03942913
Title: Real-world Prospective Registry to Describe the Current Treatment Patterns With Oral Anticoagulant and Antiplatelet Agents Association in Patients With Atrial Fibrillation and Undergoing Percutaneous Coronary Intervention
Brief Title: Prospective Real-world Registry Describing Treatment Regimens
Acronym: PRAETORIAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-20; 2019-A00325-52 (Registry Identifier: APHM)
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Subject Under Anticoagulant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dual therapy: including 1 antiplatelet treatment aspirin or clopidogrel associated with 1 anticoagulant treatment VKA or NOAC.
  Interventions: Other: an observational study
- triple therapy: including 2 antiplatelet treatments (aspirin and clopidogrel) associated with 1 anticoagulant treatment VKA or NOAC.
  In VKA class, 2 different drugs are commonly prescribed: warfarin and fluidinione. In NOAC class, 3 different drugs are commonly prescribed: rivaroxaban, apixaban, dabigatran.
  Interventions: Other: an observational study

INTERVENTIONS:
Other: an observational study — this study is to describe the initial anti-thrombotic treatment strategy prescribed to the AF patient population undergoing PCI by using drug class description.

SUMMARY:
This study is to describe the initial anti-thrombotic treatment strategy prescribed to the AF patient population undergoing PCI by using drug class description.

DETAILED DESCRIPTION:
Coordinator of project has strong expertise in cardiovascular research and especially in ACS, PCI and antiplatelet therapy. The group led by pr Bonello has published several articles (appendix 3) including the VASP studies which have been presented at major cardiologic congresses (late breaking trials ACC 2007, AHA 2008, TCT 2011, EuroPCR 2010) including physicians and biologists. The group is composed of international experts in this research field (Pr Bonello, Pr Cuisset, Dr Barragan, Pr Lemesle). Additionally, coordinator center has a strong expertise in clinical research and a methodological support will be provided by the Clinical Research Platform of the AP-HM (responsible: Prof. Pascal Auquier, medical referent: Dr Karine Baumstarck).

The project brings together investigators that have been previously involved in many clinical studies in the field of ACS and PCI. In particular they have joined forces on multicenter trials leaded by the cardiology department of the Hôpital Universitaire Nord de Marseille (the VASP studies, the Early clinical trial) and they have regular meetings to share scientific data and research program design and advancement. There is a good capacity and ability of recruitment by the partner centers. The procedures to perform in this project are very simple and the disease is frequent. These are good criteria for the feasibility.

ELIGIBILITY:
Inclusion Criteria:

The eligible subjects must meet all of the following criteria:

* Man or woman 18 years old or over
* Subject requiring percutaneous coronary intervention according to physician's and with AF requiring chronic anticoagulation by dual therapy or triple therapy;
* Subject with pulmonary embolism risk score > 1 for men and ≥ 1 for women in CHA2DS2-VASc classification
* Subject having declare its non-opposition to study participation

Exclusion Criteria:

* Child-bearing potential (1 year post-menopausal, contraceptive or surgically sterile)
* Lactation
* No health insurance
* Prisoners

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The recruiting will be performed in emergency and cardiologic units by using a consecutive screening and enrollment strategy. Information obtained as part of routine care will be reviewed to determine eligibility for enrollment including 12 lead electrocardiograms and medical exam, cardiac biomarker and all means considered necessary for diagnosis of intermediate-risk and high-risk ACS. For all patients undergoing an invasive strategy and requiring chronic anticoagulant therapy for AF, the site will carefully review the inclusion and exclusion criteria described in the protocol to confirm the subject's eligibility.
Sampling Method: Probability Sample
Enrollment: 573 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
frequency of patients treated after PCI with each drug class. | 1 year

SECONDARY OUTCOMES:
The type, the daily dosage and the duration of each drug class | 18 MONTHS
The type, the daily dosage and the duration of each drug combination | 18 MONTHS
tthe type of bleeding events according TIMI classification1 for each drug | 18 MONTHS
The major adverse cardiovascular events (MACE) | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France